CLINICAL TRIAL: NCT01336777
Title: Heterogeneity of Fat Depots
Brief Title: Regional Fat Depots and Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of California (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Tracey McLaughlin, Associate Professor, Stanford University
Other Study IDs: 1R01DK080436 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-18 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Insulin Resistance; Diabetes Mellitus Type 2
Keywords: obesity; adipocyte differentiation; inflammation; insulin resistance; visceral fat; regional fat depots
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — adipose tissue samples will be frozen for gene expression analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Insulin resistant group: there is no intervention
- Insulin sensitive group: There is no intervention

SUMMARY:
The biological basis for insulin resistance associated with obesity is unknown. By studying equally-overweight/obese individuals who are either insulin resistant or insulin sensitive, the investigators will compare characteristics of fat tissue to test several hypotheses: 1) impaired differentiation and fat storage in the subcutaneous fat depot characterize insulin resistant individuals, who have, as a result, fat in other tissues like liver and muscle, as well as more fat circulating in the blood; 2) inflammation is greater in visceral and/or subcutaneous adipose tissue depots in insulin resistant individuals as compared with insulin sensitive individuals.

DETAILED DESCRIPTION:
Insulin resistance (IR) is a major contributor to obesity-related morbidities such as diabetes and cardiovascular disease. While obesity is associated with IR, the biological basis for this association is unclear, and not all obese individuals are IR. The once-popular portal hypothesis, which states that lipolysis from VAT in particular accounts for IR, has been questioned because VAT contributes only 15% of the total systemic free fatty acid (FFA) flux. Other proposed mechanisms linking obesity to IR include inflammation, adiponectin, and ectopic fat. It is unclear whether VAT mass is more closely linked to IR than is subcutaneous adipose tissue (SAT) mass. Furthermore, evidence linking differential biological activity to IR in VAT or SAT is indirect, largely derived from studies comparing lean to obese or VAT to SAT without evaluation of IR. Thus, the purpose of this study is to investigate the biological mechanisms by which SAT and/or VAT contribute to IR. Specifically, the investigators will explore two related hypotheses- that impaired adipocyte differentiation in SAT is related to IR, ectopic fat deposition and expansion of VAT depot, and that inflammation in VAT is associated with IR. Utilizing adipose cell size/distribution obtained by Beckman Coulter Multisizer, gene expression via quantitative PCR, in-vivo quantification of IR via a modified insulin suppression test, and CT scans of abdomen/thigh, our specific aims are to:

1. Confirm that impairment of adipocyte differentiation in SAT is associated with IR by comparing cell size characteristics and differentiation markers in IR and IS subjects undergoing elective surgery;
2. Test the hypothesis that the same relationship will not be seen in VAT;
3. Demonstrate that VAT mass is expanded in the presence of impaired differentiation of adipocytes in SAT;
4. Demonstrate that intramuscular fat is related to both IR and impaired differentiation of adipocytes in SAT using cell size characteristics and differentiation markers;
5. Demonstrate that increased inflammation in omental fat is associated with IR independent of obesity using inflammation markers (gene and protein).

ELIGIBILITY:
Inclusion Criteria:

* No major organ disease
* Fasting blood glucose < 126 mg/dL
* BMI 25-35 kg/m2
* Nonpregnant/nonlactating

Exclusion Criteria:

* pregnancy/lactation
* major organ disease
* drugs that influence insulin resistance
* unstable body weight or active weight loss program
* outside BMI range or age range
* diabetic by fasting glucose criteria 126 mg/dL or higher

Ages: 39 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, nondiabetic volunteers will be recruited from Stanford's General Surgery Preoperative Clinic, Stanford's Bariatric Surgery Clinic, and nonsurgical volunteers who respond to local newspaper advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Adipose Cell Size | 3 years
  Harvest adipose tissue from human biopsy. Prepare for cell size analysis using Beckman Multisizer Coulter Counter

SECONDARY OUTCOMES:
Macrophage density | 3 years
  Human adipose tissue will be formalin-fixed and paraffin-blocked for immunohistochemical analysis to identify macrophage number and pattern
Gene Expression | 3 years
  Adipose tissue from humans will be frozen and RNA prepared for measurement of relative expression of genes related to adipose cell differentiation, fat storage, and inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] McLaughlin T, Lamendola C, Liu A, Abbasi F. Preferential fat deposition in subcutaneous versus visceral depots is associated with insulin sensitivity. J Clin Endocrinol Metab. 2011 Nov;96(11):E1756-60. doi: 10.1210/jc.2011-0615. Epub 2011 Aug 24. PMID 21865361